CLINICAL TRIAL: NCT05578859
Title: A Phase I, Open-label Study of the Absorption, Metabolism, and Excretion of [14C]-AMG 510 Following a Single Oral Dose in Healthy Male Subjects
Brief Title: A Study of the Absorption, Metabolism, and Excretion of [14C]-AMG 510 Following a Single Oral Dose in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20190321
Record Dates: First submitted 2022-10-11; First posted 2022-10-13 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Healthy Subjects
Keywords: Healthy volunteers; AMG 510
MeSH Terms: interventions — sotorasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AMG510 (Experimental): Each participant will receive a single oral dose of AMG510 on Day 1 after an overnight fast.
  Interventions: Drug: AMG 510

INTERVENTIONS:
Drug: AMG 510 — Single oral dose of AMG510.

SUMMARY:
The primary objectives of the study are: to characterize the primary route(s) of elimination of [14C]-AMG 510 and drug-related material, and estimate the overall recovery of radiolabeled material in healthy male participants after oral administration of [14C]-AMG 510, and to characterize the pharmacokinetic (PK) of total radioactivity and AMG 510 following a single oral dose of [14C]-AMG 510 in healthy male participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male participants between 18 and 55 years of age (inclusive) at the time of Screening.
* In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, and clinical laboratory evaluations as assessed by the Investigator (or designee).
* Body mass index between 18 and 30 kg/m2 (inclusive) at the time of Screening.
* History of a minimum of 1 bowel movement per day.

Exclusion Criteria:

* History or evidence, at Screening or Check-in, of clinically significant disorder, condition, or disease not otherwise excluded that, in the opinion of the Investigator (or designee), would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion.
* History suggestive of esophageal (including esophageal spasm, esophagitis), gastric, or duodenal ulceration or bowel disease (including but not limited to peptic ulceration, gastrointestinal bleeding, ulcerative colitis, Crohn's disease, or irritable bowel syndrome); or a history of gastrointestinal surgery other than uncomplicated appendectomy.
* Inability to swallow oral medication or history of malabsorption syndrome.
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee) and in consultation with the Sponsor.
* Poor peripheral venous access.
* History of alcoholism or drug/chemical abuse within 1 year prior to Check-in.
* Participant has received a dose of an investigational drug (new chemical entity) within the past 90 days or 5 half-lives, whichever is longer, prior to Check-in.
* Participants with exposure to significant diagnostic or therapeutic radiation (eg, serial X-ray, computed tomography scan, barium meal) or current employment in a job requiring radiation exposure monitoring within 12 months prior to Check-in.
* Participants who have participated in a radiolabeled drug study where exposures are known to the Investigator within the previous 4 months prior to admission to the clinic for this study or participated in a radiolabeled drug study where exposures are not known to the Investigator within the previous 6 months prior to admission to the clinic for this study. The total 12-month exposure from this study and a maximum of 2 other previous radiolabeled studies within 4 to 12 months prior to this study will be within the Code of Federal Regulations (CFR)-recommended levels considered safe, per US Title 21 CFR 361.1: less than 5000 mrem whole body annual exposure with consideration given to the half-lives of the previous radiolabeled study drugs received.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve (AUC) from time zero to infinity (AUCinf) | Day 1 to Day 14
AUC from time zero to the last quantifiable concentration (AUClast) | Day 1 to Day 14
Maximum observed concentration (Cmax) | Day 1 to Day 14
Time of Cmax (tmax) | Day 1 to Day 14
Apparent terminal elimination half-life (t1/2) | Day 1 to Day 14
Total clearance (AMG 510 only; CL/F) | Day 1 to Day 14
Volume of distribution (AMG 510 only; Vz/F) | Day 1 to Day 14
Plasma AMG 510 to total radioactivity ratio | Day 1 to Day 14
Whole blood to plasma total radioactivity ratio | Day 1 to Day 14
Amount (Aeu) of AMG510 excreted in urine | Day 1 to Day 14
Percentage (feu) of AMG510 excreted in urine | Day 1 to Day 14
Renal clearance (CLR) of AMG510 | Day 1 to Day 14
Amount (Aef) of AMG510 excreted in feces | Day 1 to Day 14
Percentage (fef) of AMG510 excreted in feces | Day 1 to Day 14

SECONDARY OUTCOMES:
Metabolite profile of AMG 510 | Day 1 to Day 14
Identification of AMG 510 metabolites | Day 1 to Day 14
Incidence of adverse events | Up to approximately 6 weeks
  Adverse events will be graded by severity. Laboratory abnormalities (hematology, clinical chemistry, and urinalysis test results) will be recorded as adverse events, in addition to abnormalities in vital signs and physical examinations.
QTc interval measured by 12-lead electrocardiogram (ECG) | Up to approximately 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Covance Clinical Research Unit, Inc, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com